CLINICAL TRIAL: NCT06746727
Title: The Development of a Transdiagnostic Intervention to Improve Social Functioning and Intimate Relationships Among Veterans
Acronym: ACT-SHARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5027-W
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Problems; Post-Traumatic Stress Disorder
Keywords: Social Functioning; Intimate Partner Abuse; Post-Traumatic Stress Disorder; Alcohol Problems; Acceptance and Commitment Therapy
MeSH Terms: conditions — Alcohol-Related Disorders; Stress Disorders, Post-Traumatic; Social Adjustment

STUDY DESIGN:
Intervention Model Description: This single-arm intervention will pilot a new, manualized intervention adapted from existing interventions using Acceptance and Commitment Therapy (ACT) to address alcohol use, PTSD, social functioning, and IPV use. ACT for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE) aims to assist Veterans in developing skills central to psychological flexibility (e.g., acceptance, mindfulness, commitment to values-based action) to improve their relationship functioning and decrease IPV use in the presence of PTSD symptoms (e.g., anger, irritability, detachment from others) and alcohol use issues (e.g., cravings, triggers, disconnection from valued roles).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACT-SHARE (Experimental): This is a single-arm intervention with all participants assigned to receive Acceptance and Commitment Therapy for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE). ACT-SHARE has been adapted for this study from existing interventions using Acceptance and Commitment Therapy (ACT) to address alcohol use, PTSD, social functioning, and IPV use.
  Interventions: Behavioral: Acceptance and Commitment Therapy for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE) — This single-arm intervention will pilot a new, manualized intervention adapted from existing interventions using Acceptance and Commitment Therapy (ACT) to address alcohol use, PTSD, social functioning, and IPV use. ACT for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE) aims to assist Veterans in developing skills central to psychological flexibility (e.g., acceptance, mindfulness, commitment to values-based action) to improve their relationship functioning and decrease IPV use in the presence of PTSD symptoms (e.g., anger, irritability, detachment from others) and alcohol use issues (e.g., cravings, triggers, disconnection from valued roles).
  Other Names: ACT-SHARE

SUMMARY:
Veterans seeking to improve their romantic relationships when high conflict and unhealthy dynamics (e.g., aggression) are present remain underserved within the VHA with few treatment options. Veterans with PTSD and alcohol misuse face compounding and overlapping barriers to intimate relationship functioning warranting tailored interventions. These Veterans may be best served through individual, Acceptance and Commitment Therapy (ACT) interventions which can both 1) improve the ability to manage challenging, internal experiences (e.g., physiological reactivity, cravings, beliefs about worth and trust) and 2) encourage participation in valued actions to improve relationship functioning. Following development and refinement, this clinical trial will pilot an evidence-based, integrated ACT intervention (ACT for Social Health, Achievement, and Relationship Effectiveness [ACT-SHARE]) to improve relationship health and safety for Veterans with PTSD alcohol misuse.

DETAILED DESCRIPTION:
Romantic partnerships greatly impact mental and physical wellness. However, these vital relationships are frequently put at risk by behaviors which put the health and safety of relationships at risk such as high interpersonal conflict or aggression (intimate partner violence [IPV]). Veterans endorse high rates of relationship conflict which frequently include the use of physical or psychological aggression toward a partner. As a prevalent and detrimental problem, interventions are gravely needed that consider primary drivers of relationship conflict and aggression: internal emotional processes and intimate relationship functioning (e.g., intimacy, communication, conflict resolution). Intervention development holds particular importance for Veterans who have few treatment options and present with distinct risk factors. For instance, co-occurring PTSD and alcohol misuse (i.e., hazardous alcohol use or alcohol use disorder; AUD) exacerbate risk for intimate relationship dysfunction and IPV use among Veterans through overlapping processes (e.g., emotional numbing, social erosion, increased threat perception). Despite high prevalence of co-occurrence and well-defined impact on relationship functioning and IPV use risk, Veterans with PTSD and alcohol misuse are not well served by couple's interventions, IPV use treatments, or evidence-based practices for co-occurring disorders. Veterans endorsing high relationship conflict, particularly when reaching the point of IPV use, are frequently excluded from services or sent to several, distinct interventions to treat intersecting problems such as alcohol misuse and PTSD. While evidenced based interventions for PTSD and alcohol misuse show distinct promise in symptom reduction, they do not necessarily improve psychosocial functioning. Relationship health and safety interventions do not yet exist which provide tailored, individual programming. With these limitations, existing referral lines for increase likelihood for dropout and evidence higher rates of poor relationship functioning and IPV following treatment. A new intervention is needed which can provide individualized treatment for Veterans with PTSD and alcohol misuse targeting intimate relationship functioning and IPV reduction. Acceptance and Commitment Therapy (ACT) is a promising avenue for intervention development. Increasing "psychological flexibility" via ACT, or value-driven functioning in the presence of challenging internal experiences, addresses a transdiagnostic process spanning across PTSD, alcohol misuse, intimate relationship functioning, and IPV use. This five year Rehabilitation Research Development and Translation (RRDT) career development award aims to develop, refine, and pilot this individual, manualized treatment called: ACT for Social Health, Achievement, and Relationship Effectiveness (ACT-SHARE). Following Phase 1 which will develop the intervention and Phase 2 which will refine the intervention through iterative feedback, Phase 3 will pilot the adapted intervention, full trial procedures including 12-month follow-up, and training and rating procedures. Primary aims include feasibility and acceptability with exploratory aims examining change scores (relationship functioning, IPV use, PTSD symptoms, alcohol use) and candidate processes (psychological flexibility).

ELIGIBILITY:
Inclusion Criteria:

* Endorses at least one act of IPV in the past 3 months
* Endorses treatment goals related to improving romantic relationship functioning
* Meets DSM 5 Criteria for PTSD and screening cutoffs for alcohol misuse (mild to severe AUD criteria met and/or above AUDIT cutoff).
* Consents to audio recording.
* Able to provide informed consent.
* Consents to partner outreach if in a relationship.
* Over 18 years of age

Exclusion Criteria:

* Evidence of active psychosis or mania
* Suicidality requiring inpatient hospitalization
* Severity of active substance use requiring detoxification
* Cognitive impairment that would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2028-07-03 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Week 12
  The CSQ-8 is a commonly used, 8-item measure to assess treatment satisfaction (administered at post-treatment and follow ups).

SECONDARY OUTCOMES:
Multidimensional Psychological Flexibility Inventory (MPFI) | Week 3, Week 12, 3-month Follow-up, 6-month Follow-up
  The MPFI, a 30-item self-report measure, assesses psychological flexibility across 6 dimensions: present moment awareness, self as context, acceptance, contact with values, committed action, cognitive defusion; and psychological inflexibility across 6 dimensions: cognitive fusion, self as context, inaction, lack of contact with values, lack of contact with the present moment, experiential avoidance, and 2 global composite scores. The MFPI is sensitive to clinical change within interventions.
Interpersonal Confidence Questionnaire (ICQ) | Week 3, Week 12, 3-month Follow-up, 6-month Follow-up
  The ICQ, a 40-item self-report measure, assesses intimate relationship functioning across 5 domains: relationship initiation, asserting displeasure, emotional disclosure, providing emotional support, and conflict management. The ICQ is a comprehensive measure of intimate relationship functioning and has demonstrated sensitivity to change in randomized controlled trials for IPV use consistent with the proposed study's follow-up points.
Revised Conflict Tactics Scales 2 Revised Short Form (CTS-2 SF) | 3-month Follow-up, 6-month Follow-up
  20 items will assess IPV use and experience in the following domains: physical assault, sexual coercion, psychological aggression, injury, and negotiation. The CTS-2 therefore assesses both the use of violence and adaptive use of non-violent conflict resolution strategies. The CTS-2 is the gold standard for IPV assessment with well-established psychometric properties including construct, convergent, and discriminant validity. The CTS-2 was developed to assess annual and lifetime IPV rates and will be adapted to the current study to assess the past 3 months.
Alcohol Use Disorders Identification Test (AUDIT) | Week 3, Week 12, 3-month Follow-up, 6-month Follow-up
  The AUDIT (10 items)assesses drinking frequency, quantity, intensity, dependence, tolerance, and consequences. Items are summed to receive a total score from 0-40. Higher scores indicate greater alcohol use and associated problems. Good reliability and validity have been demonstrated in empirical studies.5 The World Health Organization (WHO) defines scores 8-14 as "hazardous drinking" while scores 15 or above signal probable dependence.
PTSD Checklist (PCL-5) | Week 3, Week 12, 3-month Follow-up, 6-month Follow-up
  The PCL-5 is a 20-item self-report measure of PTSD symptoms. The PCL-5 is sensitive across diagnostic dimensions of PTSD with higher scores reflecting greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Grigorian, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No